CLINICAL TRIAL: NCT01513109
Title: A Phase I/II Study to Assess the Safety and Immunogenicity of WT1-A10 + AS01B Antigen-Specific Cancer Immunotherapeutic (ASCI) Combined With Infusions of ex Vivo Regulatory T Cells Depleted T Lymphocytes in in Vivo Regulatory T Cells Depleted Patients as Post-consolidation Therapy for Adult Patients With WT1-positive Acute Myeloid Leukemia (AML) in CR1 (for High Risk Patients) or in CR2 or CR3 Who Are Not Eligible for Allogeneic Stem Cell Transplantation (SCT).
Brief Title: Safety and Immunogenicity of Recombinant WT1 Antigen-Specific Cancer Immunotherapeutic Combined With Infusion of Treg Depleted T Cells for Adult WT1 Acute Myeloid Leukemia
Acronym: ASCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BORLEUWT01
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Acute Myelogenous Leukemia; Myeloid Leukemia in Remission; Effects of Immunotherapy
Keywords: WT1 positive Acute Myeloid Leukemia; Antigen specific cancer immunotherapeutic; Ex vivo regulatory T cell depletion; In vivo regulatory T cell depletion
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Recombinant WT1 Antigen-Specific Cancer Immunotherapeutic combined with Treg depletion
  Interventions: Biological: Recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI)

INTERVENTIONS:
Biological: Recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) — i.m. administration

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of combined treatment strategy of WT1ASCI, infusion of ex vivo regulatory T cells depleted T lymphocytes and in vivo regulatory T cells depletion as post-consolidation therapy in patients with WT1-positive Acute Myeloid Leukemia. The study will also evaluate the clinical activity and immune response of this approach in bad risk patients in CR1 and all patients in CR2 or CR3, non eligible for an allogeneic Hematopoietic Stem Cell Transplantation

DETAILED DESCRIPTION:
High-risk and intermediate-high risk CR1 AML patients who are not eligible for allo-SCT after chemotherapy have an unfavorable prognosis, and there is currently no treatment able to improve their survival. New approaches to treat these patients are thus urgently needed. Active immunization against tumor antigens is certainly one of these approaches. The tumor antigen targeted in this study is WT1, which is overexpressed and acts as an oncogene in leukemia and several types of solid tumors. WT1-positive acute myeloid Leukemia patients in complete remission (CR) will first undergo two cytaphereses, one of which being frozen, after CD25+ T cell depletion, the second, being frozen unmanipulated as a Treg back-up. Next, patients will be treated for 5 weeks with oral cyclophosphamide according to the so-called "metronomic regimen" to achieve in vivo Treg depletion. Patients will thereafter receive WT1 ASCI combined with CD25+ T cell depleted lymphocytes. The total duration of the treatment period will last 48 months (4 years).

ELIGIBILITY:
Inclusion Criteria:

1. The patient has cytologically proven AML, as defined by the WHO classification. The leukemia is a de novo or a secondary leukemia.
2. The patient is in complete morphologic remission Note: Cytogenetic CR (CRc) or molecular CR (CRm) is not required.

   * AML patients in first complete remission (CR1) who are not eligible for allo-HSCT following the institution's standard of care(except the favourable genetic group subset which is excluded from this study).
   * All AML patients in second or third complete morphological remission(CR2 or CR3) who are not eligible for allo-HSCT.
3. The patient received the following therapy according to the institution's standard of care:

   * For patients ≤ 60 years old, at least two cycles of intensive chemotherapy (induction and consolidation)
   * For patients > 60 years old, at least one induction chemotherapy. Any patients with severe co-morbidity for which consolidation is unacceptable, can receive only one induction therapy.
4. The patient's blasts cells show over-expression of WT1 transcripts, detected in peripheral blood by qRT-PCR at diagnosis or at first relapse.
5. Written informed consent has been obtained prior to the performance of any protocol-specific procedure.
6. The patient is ≥ 18 years of age at the time of signing of the ICF.
7. ECOG performance status of 0, 1, or 2 at the time of enrollment.
8. Adequate hepatic and renal function defined as:

   * Serum bilirubin < 1.5 times the Upper Limit of Normal (ULN).
   * Serum alanine aminotransferase ALAT < 2.5 times the ULN.
   * Calculated creatinine clearance > 40 mL/min.
9. If the patient is female, then she must be of non-childbearing potential, i.e., have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal, or if she is of childbearing potential, then she must practice adequate contraception for 30 days prior to treatment administration, have a negative pregnancy test, and continue such precautions for two months after completion of the treatment administration series.
10. Under the investigator criteria, the patient is able to comply with the protocol requirements during the duration of the study.
11. In the investigator's opinion and in compliance with the Institution hematology guidance, the patient should not be eligible for an approved standard of care such as induction with chemotherapy or allo-HSCT.

Exclusion Criteria:

1. The patient is in morphologic leukemia-free state or in morphologic complete remission but with incomplete blood count recovery as defined by IWG Response Criteria
2. The patient is in CR1 and is in the category of low-risk for relapse patients, i.e. belong to the favourable genetic group subset .
3. The patient was diagnosed with leukemic central nervous system (CNS) disease (E.g. before chemotherapy) or presents neurological symptoms at baseline suggestive of a CNS involvement.
4. The patient has received, is receiving (or is due to receive) allo-HSCT.
5. The patient has (or has had) concomitant malignancies, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
6. The patient is known to be human immunodeficiency virus (HIV)-positive.
7. The patient has symptomatic autoimmune disease such as, but not limited to, multiple sclerosis, lupus, rheumatoid arthritis and inflammatory bowel disease.
8. The patient has a history of allergic reactions likely to be exacerbated by any component of the study investigational product.
9. The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
10. The patient has congestive heart failure, symptomatic coronary artery disease, or previous myocardial infarction.
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
12. The patient has received any investigational or non-registered medicinal product other than the study medication within 30 days preceding the first dose of study medication, or plans to receive such a drug during the study period.
13. The patient requires concomitant treatment with systemic corticosteroids or any other immunosuppressive agents. The use of prednisone, or equivalent, < 0.5 mg/kg/day (absolute maximum 40 mg/day), inhaled corticosteroids or topical steroids is permitted.
14. The patient has an active infection and/or is receiving antibiotics. The patient has received i.v. administration of antibiotics within two weeks prior to first study treatment or oral antibiotics within one week prior to first study treatment.
15. For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of severe toxicities | 4 years

SECONDARY OUTCOMES:
Immunogenicity of the WT1 ASCI | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Martiat, MD PhD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, tumor center of the Universite Libre de Bruxelles, Brussels, Belgium

REFERENCES:
- [Background] Alatrash G, Molldrem JJ. Vaccines as consolidation therapy for myeloid leukemia. Expert Rev Hematol. 2011 Feb;4(1):37-50. doi: 10.1586/ehm.10.80. PMID 21322777
- [Background] Barrett AJ, Le Blanc K. Immunotherapy prospects for acute myeloid leukaemia. Clin Exp Immunol. 2010 Aug;161(2):223-32. doi: 10.1111/j.1365-2249.2010.04197.x. Epub 2010 May 31. PMID 20529084
- [Background] Cao X. Regulatory T cells and immune tolerance to tumors. Immunol Res. 2010 Mar;46(1-3):79-93. doi: 10.1007/s12026-009-8124-7. PMID 19763889
- [Background] Zhao J, Cao Y, Lei Z, Yang Z, Zhang B, Huang B. Selective depletion of CD4+CD25+Foxp3+ regulatory T cells by low-dose cyclophosphamide is explained by reduced intracellular ATP levels. Cancer Res. 2010 Jun 15;70(12):4850-8. doi: 10.1158/0008-5472.CAN-10-0283. Epub 2010 May 25. PMID 20501849
- [Background] Cao Y, Zhao J, Yang Z, Cai Z, Zhang B, Zhou Y, Shen GX, Chen X, Li S, Huang B. CD4+FOXP3+ regulatory T cell depletion by low-dose cyclophosphamide prevents recurrence in patients with large condylomata acuminata after laser therapy. Clin Immunol. 2010 Jul;136(1):21-9. doi: 10.1016/j.clim.2010.02.020. Epub 2010 Mar 24. PMID 20338811
- [Background] Casalegno-Garduno R, Schmitt A, Wang X, Xu X, Schmitt M. Wilms' tumor 1 as a novel target for immunotherapy of leukemia. Transplant Proc. 2010 Oct;42(8):3309-11. doi: 10.1016/j.transproceed.2010.07.034. PMID 20970678
- [Background] Copier J, Dalgleish AG, Britten CM, Finke LH, Gaudernack G, Gnjatic S, Kallen K, Kiessling R, Schuessler-Lenz M, Singh H, Talmadge J, Zwierzina H, Hakansson L. Improving the efficacy of cancer immunotherapy. Eur J Cancer. 2009 May;45(8):1424-31. doi: 10.1016/j.ejca.2008.12.017. Epub 2009 Jan 21. PMID 19167214
- [Background] Nizar S, Copier J, Meyer B, Bodman-Smith M, Galustian C, Kumar D, Dalgleish A. T-regulatory cell modulation: the future of cancer immunotherapy? Br J Cancer. 2009 Jun 2;100(11):1697-703. doi: 10.1038/sj.bjc.6605040. Epub 2009 Apr 21. PMID 19384299
- [Background] Dao T, Scheinberg DA. Peptide vaccines for myeloid leukaemias. Best Pract Res Clin Haematol. 2008 Sep;21(3):391-404. doi: 10.1016/j.beha.2008.05.001. PMID 18790445
- [Background] Tsuboi A, Oka Y, Kyo T, Katayama Y, Elisseeva OA, Kawakami M, Nishida S, Morimoto S, Murao A, Nakajima H, Hosen N, Oji Y, Sugiyama H. Long-term WT1 peptide vaccination for patients with acute myeloid leukemia with minimal residual disease. Leukemia. 2012 Jun;26(6):1410-3. doi: 10.1038/leu.2011.343. Epub 2011 Dec 13. No abstract available. PMID 22157809
- [Background] Tamura H, Dan K, Yokose N, Iwakiri R, Ohta M, Sakamaki H, Tohyama K, Kondo A, Hyodo H, Nakamura K, Yamashita T, Elisseeva OA, Oka Y, Oji Y, Sugiyama H, Ogata K. Prognostic significance of WT1 mRNA and anti-WT1 antibody levels in peripheral blood in patients with myelodysplastic syndromes. Leuk Res. 2010 Aug;34(8):986-90. doi: 10.1016/j.leukres.2009.11.029. Epub 2010 Jan 19. PMID 20031209
- [Background] Fujiki F, Oka Y, Kawakatsu M, Tsuboi A, Nakajima H, Elisseeva OA, Harada Y, Li Z, Tatsumi N, Kamino E, Shirakata T, Nishida S, Taniguchi Y, Kawase I, Oji Y, Sugiyama H. A WT1 protein-derived, naturally processed 16-mer peptide, WT1(332), is a promiscuous helper peptide for induction of WT1-specific Th1-type CD4(+) T cells. Microbiol Immunol. 2008 Dec;52(12):591-600. doi: 10.1111/j.1348-0421.2008.00080.x. PMID 19120973
- [Background] Elisseeva OA, Oka Y, Tsuboi A, Ogata K, Wu F, Kim EH, Soma T, Tamaki H, Kawakami M, Oji Y, Hosen N, Kubota T, Nakagawa M, Yamagami T, Hiraoka A, Tsukaguchi M, Udaka K, Ogawa H, Kishimoto T, Nomura T, Sugiyama H. Humoral immune responses against Wilms tumor gene WT1 product in patients with hematopoietic malignancies. Blood. 2002 May 1;99(9):3272-9. doi: 10.1182/blood.v99.9.3272. PMID 11964293
- [Background] Elkord E, Alcantar-Orozco EM, Dovedi SJ, Tran DQ, Hawkins RE, Gilham DE. T regulatory cells in cancer: recent advances and therapeutic potential. Expert Opin Biol Ther. 2010 Nov;10(11):1573-86. doi: 10.1517/14712598.2010.529126. PMID 20955112
- [Background] Fujiki F, Oka Y, Kawakatsu M, Tsuboi A, Tanaka-Harada Y, Hosen N, Nishida S, Shirakata T, Nakajima H, Tatsumi N, Hashimoto N, Taguchi T, Ueda S, Nonomura N, Takeda Y, Ito T, Myoui A, Izumoto S, Maruno M, Yoshimine T, Noguchi S, Okuyama A, Kawase I, Oji Y, Sugiyama H. A clear correlation between WT1-specific Th response and clinical response in WT1 CTL epitope vaccination. Anticancer Res. 2010 Jun;30(6):2247-54. PMID 20651376
- [Background] Ghiringhelli F, Menard C, Puig PE, Ladoire S, Roux S, Martin F, Solary E, Le Cesne A, Zitvogel L, Chauffert B. Metronomic cyclophosphamide regimen selectively depletes CD4+CD25+ regulatory T cells and restores T and NK effector functions in end stage cancer patients. Cancer Immunol Immunother. 2007 May;56(5):641-8. doi: 10.1007/s00262-006-0225-8. Epub 2006 Sep 8. PMID 16960692
- [Background] Golovina TN, Vonderheide RH. Regulatory T cells: overcoming suppression of T-cell immunity. Cancer J. 2010 Jul-Aug;16(4):342-7. doi: 10.1097/PPO.0b013e3181eb336d. PMID 20693845
- [Background] Ochsenreither S, Fusi A, Busse A, Bauer S, Scheibenbogen C, Stather D, Thiel E, Keilholz U, Letsch A. "Wilms Tumor Protein 1" (WT1) peptide vaccination-induced complete remission in a patient with acute myeloid leukemia is accompanied by the emergence of a predominant T-cell clone both in blood and bone marrow. J Immunother. 2011 Jan;34(1):85-91. doi: 10.1097/CJI.0b013e3181f3cc5c. PMID 21150716
- [Background] Keilholz U, Letsch A, Busse A, Asemissen AM, Bauer S, Blau IW, Hofmann WK, Uharek L, Thiel E, Scheibenbogen C. A clinical and immunologic phase 2 trial of Wilms tumor gene product 1 (WT1) peptide vaccination in patients with AML and MDS. Blood. 2009 Jun 25;113(26):6541-8. doi: 10.1182/blood-2009-02-202598. Epub 2009 Apr 23. PMID 19389880
- [Background] Maslak PG, Dao T, Krug LM, Chanel S, Korontsvit T, Zakhaleva V, Zhang R, Wolchok JD, Yuan J, Pinilla-Ibarz J, Berman E, Weiss M, Jurcic J, Frattini MG, Scheinberg DA. Vaccination with synthetic analog peptides derived from WT1 oncoprotein induces T-cell responses in patients with complete remission from acute myeloid leukemia. Blood. 2010 Jul 15;116(2):171-9. doi: 10.1182/blood-2009-10-250993. Epub 2010 Apr 16. PMID 20400682
- [Background] Mougiakakos D, Choudhury A, Lladser A, Kiessling R, Johansson CC. Regulatory T cells in cancer. Adv Cancer Res. 2010;107:57-117. doi: 10.1016/S0065-230X(10)07003-X. PMID 20399961
- [Background] Nakahara T, Uchi H, Lesokhin AM, Avogadri F, Rizzuto GA, Hirschhorn-Cymerman D, Panageas KS, Merghoub T, Wolchok JD, Houghton AN. Cyclophosphamide enhances immunity by modulating the balance of dendritic cell subsets in lymphoid organs. Blood. 2010 Jun 3;115(22):4384-92. doi: 10.1182/blood-2009-11-251231. Epub 2010 Feb 12. PMID 20154220
- [Background] Nishikawa H, Sakaguchi S. Regulatory T cells in tumor immunity. Int J Cancer. 2010 Aug 15;127(4):759-67. doi: 10.1002/ijc.25429. PMID 20518016
- [Background] Millar MR, MacKay P, Levene M, Langdale V, Martin C. Enterobacteriaceae and neonatal necrotising enterocolitis. Arch Dis Child. 1992 Jan;67(1 Spec No):53-6. doi: 10.1136/adc.67.1_spec_no.53. PMID 1536588
- [Background] Oka Y, Sugiyama H. WT1 peptide vaccine, one of the most promising cancer vaccines: its present status and the future prospects. Immunotherapy. 2010 Sep;2(5):591-4. doi: 10.2217/imt.10.58. No abstract available. PMID 20874639
- [Background] Radojcic V, Bezak KB, Skarica M, Pletneva MA, Yoshimura K, Schulick RD, Luznik L. Cyclophosphamide resets dendritic cell homeostasis and enhances antitumor immunity through effects that extend beyond regulatory T cell elimination. Cancer Immunol Immunother. 2010 Jan;59(1):137-48. doi: 10.1007/s00262-009-0734-3. Epub 2009 Jul 10. PMID 19590872
- [Background] Rezvani K. Peptide vaccine therapy for leukemia. Int J Hematol. 2011 Mar;93(3):274-280. doi: 10.1007/s12185-011-0781-3. Epub 2011 Mar 8. PMID 21380929
- [Background] Sakaguchi S. Regulatory T cells: history and perspective. Methods Mol Biol. 2011;707:3-17. doi: 10.1007/978-1-61737-979-6_1. PMID 21287325
- [Background] Schabowsky RH, Madireddi S, Sharma R, Yolcu ES, Shirwan H. Targeting CD4+CD25+FoxP3+ regulatory T-cells for the augmentation of cancer immunotherapy. Curr Opin Investig Drugs. 2007 Dec;8(12):1002-8. PMID 18058571
- [Background] Schreiber RD, Old LJ, Smyth MJ. Cancer immunoediting: integrating immunity's roles in cancer suppression and promotion. Science. 2011 Mar 25;331(6024):1565-70. doi: 10.1126/science.1203486. PMID 21436444
- [Background] Sistigu A, Viaud S, Chaput N, Bracci L, Proietti E, Zitvogel L. Immunomodulatory effects of cyclophosphamide and implementations for vaccine design. Semin Immunopathol. 2011 Jul;33(4):369-83. doi: 10.1007/s00281-011-0245-0. Epub 2011 May 25. PMID 21611872
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Wang X, Zheng J, Liu J, Yao J, He Y, Li X, Yu J, Yang J, Liu Z, Huang S. Increased population of CD4(+)CD25(high), regulatory T cells with their higher apoptotic and proliferating status in peripheral blood of acute myeloid leukemia patients. Eur J Haematol. 2005 Dec;75(6):468-76. doi: 10.1111/j.1600-0609.2005.00537.x. PMID 16313258
- [Background] Wrzesinski C, Paulos CM, Kaiser A, Muranski P, Palmer DC, Gattinoni L, Yu Z, Rosenberg SA, Restifo NP. Increased intensity lymphodepletion enhances tumor treatment efficacy of adoptively transferred tumor-specific T cells. J Immunother. 2010 Jan;33(1):1-7. doi: 10.1097/CJI.0b013e3181b88ffc. PMID 19952961